CLINICAL TRIAL: NCT05802225
Title: A Double-Blind, Randomized Clinical Study of the Efficacy and Safety of BCD-178 and Perjeta® as Neoadjuvant Therapy of HER2-Positive Breast Cancer
Brief Title: Clinical Study of the Efficacy and Safety of BCD-178 and Perjeta® as Neoadjuvant Therapy of HER2-Positive Breast Cancer
Acronym: PREFER
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Biocad (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BCD-178-2
Record Dates: First submitted 2023-02-13; First posted 2023-04-06 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — pertuzumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- BCD-178 group (Experimental): Neoadjuvant therapy stage (6 cycles, 18 weeks): BCD-178, Trastuzumab, Docetaxel, Carboplatin; Surgical treatment; Adjuvant therapy stage (up to 12 months of HER2-targeted therapy in total): BCD-178, Trastuzumab
  Interventions: Drug: BCD-178
- Perjeta Group (Active Comparator): Neoadjuvant therapy stage (6 cycles, 18 weeks): Perjeta, Trastuzumab, Docetaxel, Carboplatin; Surgical treatment; Adjuvant therapy stage (up to 12 months of HER2-targeted therapy in total): BCD-178, Trastuzumab
  Interventions: Drug: Perjeta

INTERVENTIONS:
Drug: BCD-178 — at an initial dose of 840 mg (1 cycle), then 420 mg
  Other Names: pertuzumab
  Arms: BCD-178 group
Drug: Perjeta — at an initial dose of 840 mg (1 cycle), then 420 mg
  Other Names: pertuzumab
  Arms: Perjeta Group

SUMMARY:
The goal of this study is to compare the efficacy and safety of BCD-178 and Perjeta as neoadjuvant therapy for HER2-positive breast cancer.

Subjects with histologically confirmed diagnosis of HER2-positive invasive breast cancer (stage II-III, tumor size > 2 cm), with no estrogen (ER) and progesterone (PR) receptors will be randomized to one of two treatment groups (BCD-178 group or Perjeta group) in a 1:1 ratio.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent ;
* Histologically confirmed diagnosis of invasive breast cancer;
* Disease stage cT2-cT4, cN0-cN3, cM0;
* Positive HER2 expression, negative estrogen and progesterone receptor expression;
* ECOG score 0-1;
* Adequate organ function;
* Baseline LVEF ≥ 55%, as measured with the standard procedure;
* Consent of women of childbearing potential to use highly effective methods of contraception, starting from the signing of the informed consent form, throughout the study and for 6 months after receiving the last dose of the product.

Exclusion Criteria:

* Stage IV (metastatic) breast cancer;
* A history of any systemic therapy for breast cancer;
* Concomitant diseases and/or conditions that significantly increase the risk of adverse events during the study;
* Pregnancy or breastfeeding, as well as pregnancy planning throughout the study and for 6 months after receiving the last dose of the product;
* Hypersensitivity or allergy to any of the components of BCD-178, Perjeta, trastuzumab, carboplatin, and docetaxel.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 398 (Actual)
Dates: Start 2023-01-30 (Actual); Primary Completion 2025-06-06 (Actual); Study Completion 2026-02-20 (Estimated)

PRIMARY OUTCOMES:
To compare the efficacy of BCD-178 and Perjeta as neoadjuvant therapy by studying the total pathological complete response (tpCR) rate | immediately after the surgery
  Proportion of subjects achieving tpCR

SECONDARY OUTCOMES:
breast pathological complete response (bpCR) rate | immediately after the surgery
  Proportion of subjects achieving bpCR;
overall response rate (ORR) | at Week 18
  the ORR according to RECIST 1.1 criteria
breast-conserving surgery rate | immediately after surgery
  Proportion of subjects with breast-conserving surgery
safety assessment | up to 65 weeks
  Proportion of subjects with adverse reactions; Proportion of subjects with CTCAE 5.0 grade 3 or higher adverse reactions; • Proportion of subjects with serious adverse reactions; • Proportion of subjects who prematurely discontinued neoadjuvant therapy due to adverse reactions
immunogenicity assessment | pre-dose to week 52, 5 timepoints
  Proportion of subjects with binding and neutralizing antibodies
Pharmacokinetics assessment | pre-dose to week 18, 12 timepoints
  Cmin - minimum observed product concentration ; Ceoi - concentration at the end of each infusion

CONTACTS AND LOCATIONS:
Locations (3):
- Russia (3):
  - JSC "Modern Medical Technologies", Saint Petersburg, Sankt-Peterburg
  - The Loginov Moscow Clinical Scientific Center MHD, Moscow
  - Budgetary healthcare institution of the Omsk region "Clinical oncological dispensary", Omsk

IPD SHARING:
Plan to Share IPD: No